CLINICAL TRIAL: NCT06728605
Title: Protective Effect of Enhanced External Counterpulsation Against Negative Inflammatory Response and Organ Dysfunction After Cardiovascular Surgery
Brief Title: Protective Effect of EECP Against Negative Inflammatory Response and Organ Dysfunction After Cardiovascular Surgery
Acronym: PANDA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing Medical University (Other)
Collaborators: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Hong Liu, Principal Investigator of Department of Cardiovascular Surgery, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PANDA IX
Record Dates: First submitted 2024-12-06; First posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Coronary Heart Disease (CHD); Cardio-pulmonary Bypass; Congestive Heart Failure Chronic; Cardiogenic Shock Acute
Keywords: cardiac surgery; cardiopulmonary bypass; cardiogenic shock
MeSH Terms: conditions — Coronary Disease; Shock, Cardiogenic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- EECP group (Experimental): Patients randomly assigned to EECP received 3 half-h sessions of EECP for 3 days before surgery. Three pneumatic cuffs will be placed around the lower limbs and buttocks and will be inflated sequentially upward at the onset of diastole, and released rapidly and simultaneously before the onset of systole. The protocol-specified applied pressure will be 300 mm Hg and will be reached within 5 min of the initiation of treatment. Pulse oximetry will be monitored continuously during the treatment session, and the subject's clinical status will be re-evaluated if the oxygen saturation dropps by 4%.
  Interventions: Device: Enhanced External Counterpulsation (EECP)
- Control group (Sham Comparator): Patients randomly assigned to control received 3 half-h sessions of sham for 3 days before surgery. Three pneumatic cuffs will be placed around the lower limbs and buttocks and will be inflated sequentially upward at the onset of diastole, and released rapidly and simultaneously before the onset of systole. The protocol-specified applied pressure will be 70 mm Hg and will be reached within 5 min of the initiation of treatment. Pulse oximetry will be monitored continuously during the treatment session, and the subject's clinical status will be re-evaluated if the oxygen saturation dropps by 4%.
  Interventions: Device: Sham Comparator

INTERVENTIONS:
Device: Enhanced External Counterpulsation (EECP) — Patients randomly assigned to EECP received 3 1/2-h sessions of EECP for 3 days before surgery. Three pneumatic cuffs will be placed around the lower limbs and buttocks and will be inflated sequentially upward at the onset of diastole, and released rapidly and simultaneously before the onset of systole. The protocol-specified applied pressure will be 300 mm Hg and was reached within 5 min of the initiation of treatment. Pulse oximetry will be monitored continuously during the treatment session, and the subject's clinical status will be re-evaluated if the oxygen saturation drops by 4%.
  Arms: EECP group
Device: Sham Comparator — Patients randomly assigned to sham group received 3 1/2-h sessions of sham treatment for 3 days before surgery. Three pneumatic cuffs will be placed around the lower limbs and buttocks and will be inflated sequentially upward at the onset of diastole, and released rapidly and simultaneously before the onset of systole. The protocol-specified applied pressure will be 70 mm Hg and was reached within 5 min of the initiation of treatment. Pulse oximetry will be monitored continuously during the treatment session, and the subject's clinical status will be re-evaluated if the oxygen saturation drops by 4%.
  Arms: Control group

SUMMARY:
Enhanced external counterpulsation (EECP) is a noninvasive, non-pharmacologic intervention proven to increase nitric oxide bioavailability in patients with coronary artery disease. Although EECP showed short-term effects in improving coronary flow in patients with coronary slow flow, whether such improvement is durable remains uncertain, and the relationships between such improvement and changes in multiple organ functions as well as inflammatory markers have not been elucidated. The purpose of this study will be to evaluate the potential clinical benefits of EECP on organ function and proinflammatory cytokine concentrations during post-acute sequela of cardiovascular surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years;
* Patients with Stable angina pectoris, unstable angina pectoris, acute myocardial infarction, congestive heart failure, cardiogenic shock;
* Patients chronic heart failure;
* Patients are ready to received cardiovascular surgery during this hospital admission.
* Patients agree to participate in the study and sign an informed consent form.

Exclusion Criteria:

1. Moderate to severe aortic insufficiency; 2. Dissection aneurysm; 3. Significant pulmonary hypertension; 4, A variety of bleeding diseases or bleeding tendencies, or use anticoagulants, INR>2.0; 5, active phlebitis, venous thrombosis; 6. There is an infection in the counterpulsating limb; 7. Uncontrolled hyperhypertension (>170/110mmHg); 8. Uncontrolled arrhythmias: frequent premature beats, rapid atrial fibrillation, etc.

9. Pregnancy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
SOFA score | within the prior 7 days after cardiac surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Jun-jie Du, MD, Study Director — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Masuda D, Nohara R, Hirai T, Kataoka K, Chen LG, Hosokawa R, Inubushi M, Tadamura E, Fujita M, Sasayama S. Enhanced external counterpulsation improved myocardial perfusion and coronary flow reserve in patients with chronic stable angina; evaluation by(13)N-ammonia positron emission tomography. Eur Heart J. 2001 Aug;22(16):1451-8. doi: 10.1053/euhj.2000.2545. PMID 11482918
- [Background] Kiernan TJ, Boilson BA, Tesmer L, Harbuzariu A, Simari RD, Barsness GW. Effect of enhanced external counterpulsation on circulating CD34+ progenitor cell subsets. Int J Cardiol. 2011 Dec 1;153(2):202-6. doi: 10.1016/j.ijcard.2010.08.020. Epub 2010 Sep 16. PMID 20843569
- [Background] Sardina PD, Martin JS, Dzieza WK, Braith RW. Enhanced external counterpulsation (EECP) decreases advanced glycation end products and proinflammatory cytokines in patients with non-insulin-dependent type II diabetes mellitus for up to 6 months following treatment. Acta Diabetol. 2016 Oct;53(5):753-60. doi: 10.1007/s00592-016-0869-6. Epub 2016 Jun 9. PMID 27278477